CLINICAL TRIAL: NCT01216644
Title: A Randomized Multicenter Phase II/III Study Comparing 5-FU, Leucovorin, Oxaliplatin and Docetaxel (FLOT) Versus Epirubicin, Cisplatin and 5-FU (ECF) in Patients With Locally Advanced Resectable Adenocarcinoma of the Esophagogastreal Junction or the Stomach
Brief Title: 5-FU, Leucovorin, Oxaliplatin and Docetaxel (FLOT) Versus Epirubicin, Cisplatin and 5-FU (ECF) in Patients With Locally Advanced, Resectable Gastric Cancer
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Krankenhaus Nordwest (Other)
Responsible Party: Principal Investigator, Prof. Dr. S.E. Al-Batran, Principal Investigator, Krankenhaus Nordwest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLOT4
Record Dates: First submitted 2010-06-30; First posted 2010-10-07 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; perioperative; FLOT; ECF; pathological complete remission; locally advanced resectable adenocarcinoma of the esophagogastric juction or the stomach
MeSH Terms: conditions — Stomach Neoplasms; Pathologic Complete Response | interventions — Fluorouracil; Leucovorin; Oxaliplatin; Docetaxel; Epirubicin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FLOT (Experimental): Docetaxel 50mg/m2, d1 5-FU 2600 mg/m², d1 Leucovorin 200 mg/m², d1 Oxaliplatin 85 mg/m², d1 every two weeks (q2w) 4 cycles (8 weeks) pre-OP and 4 cycles (8 weeks) post-OP
  Interventions: Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin; Drug: Docetaxel
- ECF (Active Comparator): Epirubicin 50 mg/m2, d1 Cisplatin 60 mg/m², d1 5-FU 200 mg/m², d1-d21 every 3 weeks (q3w) 3 cycles (9 weeks) pre-OP and 3 cycles (9 weeks) post-OP
  Interventions: Drug: Epirubicin; Drug: Cisplatin; Drug: 5-fluorouracil

INTERVENTIONS:
Drug: 5-Fluorouracil — 2600 mg/m²d1 i.v. every 2 weeks
  Arms: FLOT
Drug: Leucovorin — 200 mg/m², d1, i.v., every 2 weeks
  Arms: FLOT
Drug: Oxaliplatin — 85 mg/m², d1, i.v., every 2 weeks
  Arms: FLOT
Drug: Docetaxel — 50mg/m2, d1, i.v., every 2 weeks
  Arms: FLOT
Drug: Epirubicin — 50 mg/m2, d1, i.v., every 3 weeks
  Arms: ECF
Drug: Cisplatin — 60 mg/m², d1, i.v., every 3 weeks
  Arms: ECF
Drug: 5-fluorouracil — 200 mg/m², d1-d21, i.v., every 3 weeks
  Arms: ECF

SUMMARY:
Patients with locally advanced resectable adenocarcinoma of the stomach or the esophagogastreal junction without previous therapy will be treated with one of two chemotherapy combinations before and after surgery. One half of the patients gets 5-Fluorouracil (5-FU), Leucovorin, Oxaliplatin and Docetaxel (FLOT), the others Epirubicin, Cisplatin and 5-FU (ECF). Main objective of the study is median overall survival.

DETAILED DESCRIPTION:
714 Patients with locally advanced resectable (T2-4 and/or N+, M0) adenocarcinoma of the stomach or the esophagogastreal junction without previous therapy will be included in this study. After randomization patients receive perioperatively 4 cycles FLOT or 3 cycles ECF, followed by a restaging of the tumour status and surgery. Subsequently another 4 cycles of FLOT or 3 cycles ECF are applicated. Then a central validation of the pathological remission rate is scheduled. Primary endpoint is overall survival, secondary endpoints are disease free survival, perioperative morbidity and mortality, histopathologic regression rate and R0-resection rate.

ELIGIBILITY:
Inclusion Criteria:

1. locally advanced (>T1) and/or nodal positive (N+) histologically proven adenocarcinoma of the esophagogastreal junction (AEG I-III) or the stomach without distant metastases (M0) and without infiltration of adjacent structures and organs
2. no previous surgical resection
3. no previous cytostatic chemotherapy
4. Age > 18 years (female and male)
5. ECOG ≤ 2
6. surgical resectability
7. Exclusion of peritoneal carcinomatosis (if clinically suspected) via laparoscopy
8. Leucocytes > 3.000/µl
9. Platelets > 100.000/µl
10. Serum creatinin ≤ 1.5x of normal value, or Creatinin-Clearance > 50 ml/min
11. written informed consent.
12. Ejection fraction > 50% in echocardiography before start of therapy

Exclusion Criteria:

1. distant metastases or infiltration of adjacent structures or organs and all primarily not resectable stages
2. relapse
3. Hypersensitivity against 5- Fluorouracil, Leucovorin, Oxaliplatin, Cisplatin. Epirubicin and Docetaxel
4. Existence of contraindications against 5- Fluorouracil, Leucovorin, Oxaliplatin, Cisplatin, Epirubicin or Docetaxel
5. Active CHD, Cardiomyopathy or cardiac insufficiency stage III-IV according to NYHA
6. malignant secondary disease, dated back < 5 years (exception: In-situ-carcinoma of the cervix uteri, adequately treated skin basal cell carcinoma)
7. severe non-surgical accompanying disease or acute infection
8. peripheral polyneuropathy > NCI Grad II
9. severe liver dysfunction (AST/ALT>3,5xULN, AP>6xULN, Bilirubin>1,5xULN)
10. chronic inflammable gastro-intestinal disease
11. inclusion in another clinical trial
12. pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 716 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
median overall survival | 2 years follow-up

SECONDARY OUTCOMES:
histopathological regression rate | 6 weeks after surgery
disease free survival (DFS) | 2 years follow-up
correlation of pCR and DFS with survival | 2 years follow-up
Perioperative Morbidity and Mortality | up to 2 months after surgery
R0-Resection rate | 2 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Salah-Eddin Al-Batran, MD, Principal Investigator — Institute of Clinical Cancer Research (IKF), UCT - University Cancer Center, Frankfurt, Germany
Locations (1):
- Krankenhaus Nordwest, Frankfurt, Germany

REFERENCES:
- [Derived] Zeng H, Wang C, Song LY, Jia SJ, Zeng X, Liu Q. Economic evaluation of FLOT and ECF/ECX perioperative chemotherapy in patients with resectable gastric or gastro-oesophageal junction adenocarcinoma. BMJ Open. 2022 Nov 14;12(11):e060983. doi: 10.1136/bmjopen-2022-060983. PMID 36375981
- [Derived] Koch C, Reitz C, Schreckenbach T, Eichler K, Filmann N, Al-Batran SE, Gotze T, Zeuzem S, Bechstein WO, Kraus T, Bojunga J, Dux M, Trojan J, Blumenstein I. Sarcopenia as a prognostic factor for survival in patients with locally advanced gastroesophageal adenocarcinoma. PLoS One. 2019 Oct 22;14(10):e0223613. doi: 10.1371/journal.pone.0223613. eCollection 2019. PMID 31639132
- [Derived] Al-Batran SE, Homann N, Pauligk C, Goetze TO, Meiler J, Kasper S, Kopp HG, Mayer F, Haag GM, Luley K, Lindig U, Schmiegel W, Pohl M, Stoehlmacher J, Folprecht G, Probst S, Prasnikar N, Fischbach W, Mahlberg R, Trojan J, Koenigsmann M, Martens UM, Thuss-Patience P, Egger M, Block A, Heinemann V, Illerhaus G, Moehler M, Schenk M, Kullmann F, Behringer DM, Heike M, Pink D, Teschendorf C, Lohr C, Bernhard H, Schuch G, Rethwisch V, von Weikersthal LF, Hartmann JT, Kneba M, Daum S, Schulmann K, Weniger J, Belle S, Gaiser T, Oduncu FS, Guntner M, Hozaeel W, Reichart A, Jager E, Kraus T, Monig S, Bechstein WO, Schuler M, Schmalenberg H, Hofheinz RD; FLOT4-AIO Investigators. Perioperative chemotherapy with fluorouracil plus leucovorin, oxaliplatin, and docetaxel versus fluorouracil or capecitabine plus cisplatin and epirubicin for locally advanced, resectable gastric or gastro-oesophageal junction adenocarcinoma (FLOT4): a randomised, phase 2/3 trial. Lancet. 2019 May 11;393(10184):1948-1957. doi: 10.1016/S0140-6736(18)32557-1. Epub 2019 Apr 11. PMID 30982686
- [Derived] Al-Batran SE, Hofheinz RD, Pauligk C, Kopp HG, Haag GM, Luley KB, Meiler J, Homann N, Lorenzen S, Schmalenberg H, Probst S, Koenigsmann M, Egger M, Prasnikar N, Caca K, Trojan J, Martens UM, Block A, Fischbach W, Mahlberg R, Clemens M, Illerhaus G, Zirlik K, Behringer DM, Schmiegel W, Pohl M, Heike M, Ronellenfitsch U, Schuler M, Bechstein WO, Konigsrainer A, Gaiser T, Schirmacher P, Hozaeel W, Reichart A, Goetze TO, Sievert M, Jager E, Monig S, Tannapfel A. Histopathological regression after neoadjuvant docetaxel, oxaliplatin, fluorouracil, and leucovorin versus epirubicin, cisplatin, and fluorouracil or capecitabine in patients with resectable gastric or gastro-oesophageal junction adenocarcinoma (FLOT4-AIO): results from the phase 2 part of a multicentre, open-label, randomised phase 2/3 trial. Lancet Oncol. 2016 Dec;17(12):1697-1708. doi: 10.1016/S1470-2045(16)30531-9. Epub 2016 Oct 22. PMID 27776843
- [Derived] Lorenzen S, Thuss-Patience P, Al-Batran SE, Lordick F, Haller B, Schuster T, Pauligk C, Luley K, Bichev D, Schumacher G, Homann N. Impact of pathologic complete response on disease-free survival in patients with esophagogastric adenocarcinoma receiving preoperative docetaxel-based chemotherapy. Ann Oncol. 2013 Aug;24(8):2068-73. doi: 10.1093/annonc/mdt141. Epub 2013 Apr 16. PMID 23592699